CLINICAL TRIAL: NCT03492450
Title: Unraveling Early Walking Dysfunction in Non-disabled MS People: Clinical and Instrumental Assessment of Disease Progression and Potential Therapeutic Interventions
Brief Title: Unraveling Early Walking Dysfunction in Non-disabled MS People: Assessment and Potential Therapeutic Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FISM Call 2016 cod. 2016/R/1
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2018-10

CONDITIONS: Multiple Sclerosis
Keywords: Treadmill training; Instrumented assessment; Disease progression
MeSH Terms: conditions — Multiple Sclerosis; Disease Progression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): All subjects continue participating in their normal daily and physical activities.
- Treadmill training Group (Experimental): 16 sessions (2 sessions/week for 8 weeks) of treadmill training as recommended in a review on this subject (Langeskov-Christensen, 2015) aimed at the reduction/stabilization of gait and balance disturbances.
  Interventions: Other: Treadmill training

INTERVENTIONS:
Other: Treadmill training — Tailored treatment comprising of: 1) aerobic exercises with the aim of increasing fitness 2) task-oriented balance exercises on the treadmill to improve balance and 3) cognitive behavioral interventions to improve balance and gait during dual task activities.In accordance with the literature (Langeskov-Christensen, 2015, Latimer-Cheung, 2013) the treadmill training will be carried out without body weight support, but the participants will be allowed to use the handrails for balance support if needed. The training consists of three different walking sessions, each lasting for 10 minutes: 1) preferred walking speed at an increased slope; 2) walking doing dynamic balance exercises (for example walking with feet in tandem) 3) fast gait speed defined as a 10% increase in walking speed relative to preferred speed with dual task exercises. During the 8-week intervention, walking speed in session 3 will be gradually increased with 10% to 40% of preferred speed.
  Arms: Treadmill training Group

SUMMARY:
The aim of the study is to set up a pilot study to investigate the effects of treadmill training in preventing the onset and worsening of walking impairments, balance deficits and fatigue.

DETAILED DESCRIPTION:
As regards the of potential impact of exercises on functional decline at best of our knowledge no studies have been done on preventive interventions on walking, balance and fatigue disorders in early diagnosed PwMS. However, preliminary studies found that walking exercises can improve performances in PwMS with mild disability. van der Berg et al (van der Berg, 2006) investigated whether four weeks of aerobic treadmill training would improve mobility and fatigue in PwMS. They found that aerobic treadmill training is feasible and well tolerated and walking speed and endurance increased after training without changes in reported fatigue. In agreement with this study, Sabapathy et al (Sabapathy, 2011) reported improvements in mobility after endurance exercise training. Recent reviews (Dalgas, 2008 and Heine, 2015) and a recent paper by Sandroff et al (Sandroff, 2015) suggested that endurance training at low moderate intensity is well tolerated, has beneficial effects and reduces level of fatigue in MS patients having EDSS lower than 7.

Furthermore, the long-term effects of walking based aerobic endurance exercise on gait parameters were investigated by Wonnemberg et al (Wonnemberg, 2015). They found that step cadence decreased significantly and the step length increased significantly after 12 months suggesting that walking based aerobic endurance exercise may contribute to improved gait parameters in MS patients.

Walking exercises can be performed using treadmills. A Systematic review by Swinnen et al. (Swinnen, 2012) addresses the effect of different treadmill training (TT) modalities in PwMS. It showed that treadmill training improves walking skills and distance. In addition, Braendvik et al (Braendvik, 2015) revealed that TT was superior progressive strength training in improving walking in mild to moderate PwMS. Peruzzi et al. (Peruzzi, 2016) found similar results using Virtual Reality-based TT in PwMS with mild to moderate disability. After training, gait speed, stride length and the ability in negotiating obstacles were improved. Finally Gervasoni et al (Gervasoni, 2013) showed that 3-week of treadmill training reduced fatigue in PwMS.

The Hypothesis to be tested is that treadmill training can reduce subtle balance and gait impairments decreasing the impact of MS on the activities of daily living and, thereby, favorably impact on the disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Included will be patients residing in the centers' catchment areas
* Diagnosis of Multiple Sclerosis (Polman criteria)
* Stable disease course without worsening more than 1 Expanded Disability Status Scale (EDSS) point over the last 3 months
* EDSS < 2.5,
* Disease duration shorter than or equal to 5 years,
* Releasing a written informed consent.

Exclusion Criteria:

* Multiple Sclerosis relapse within the previous three months
* Cognitive impairment (MMSE score <27);
* Diagnosis of major depression (DSM-IV);
* Severe joint and/or bone disorders interfering with balance and gait (based upon clinical judgment);
* Cardiovascular diseases;
* Unconfirmed or uncertain diagnosis of MS (Polman criteria)
* Other concomitant neurological diseases;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-12 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Change in Six Minutes Walking Test | Change from Baseline 6 minutes walking test scores at 8 weeks
  Tool used to assess walking endurance
Change in Instrumented variables | Change from Baseline scores at 8 weeks
  Gait asymmetry, Root mean squared of trunk Jerk and gait regularity on the vertical and medio-lateral plane estimated by autocorrelation coefficients (Moe-Nilssen, 2004) during the Six minutes walking test.

SECONDARY OUTCOMES:
the Twelve-Item Walking Scale | Change from Baseline Twelve-Item Walking Scale scores at 8 weeks
  Patient reported outcome about walking
the Twentyfive-foot walking test | Change from Baseline Twentyfive-foot walking test scores at 8 weeks
  Tool used to assess walking velocity
The Fatigue Severity Scale | Change from Baseline Fatigue Severity Scale scores at 8 weeks
  Patient reported outcome about fatigue
the Nine hole peg test | Change from Baseline Nine Hole Peg test scores at 8 weeks
  Tool used to assess manual dexterity

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Don Gnocchi Irccs, Milan, Italy